CLINICAL TRIAL: NCT06832631
Title: A Prospective PMCF Study of Paclitaxel Drug-coated Balloon Angioplasty for the Treatment of Symptomatic Peripheral Arterial Disease
Brief Title: VITUS Post-Market Registry
Status: Recruiting | Type: Observational
Sponsor: OrbusNeich (Industry)
Collaborators: Eucatech AG (Industry); Centre Européen de Recherche Cardiovasculaire (Unknown)
Responsible Party: Sponsor
Other Study IDs: DVAL-PLAN-064
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Arterial Disease; Peripheral Arterial Occlusive Disease
Keywords: Peripheral Arterial Disease (PAD); Peripheral Disease; Percutaneous Transluminal Angioplasty (PTA); Drug-Coated Balloon; Drug-Coated Catheter; Drug Coated Balloon (DCB)
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Arterial Occlusive Disease 1 | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VITUS peripheral drug-coated dilatation catheter: The VITUS peripheral drug-coated dilatation catheter is indicated for use in patients with peripheral arterial occlusive disease (PAOD).
  Interventions: Device: Percutaneous Transluminal Angioplasty with a paclitaxel drug-coated balloon

INTERVENTIONS:
Device: Percutaneous Transluminal Angioplasty with a paclitaxel drug-coated balloon — Balloon angioplasty for the treatment of symptomatic peripheral arterial disease with a paclitaxel drug-coated balloon

SUMMARY:
To collect post marketing surveillance data on consecutive patients with peripheral arterial occlusive disease (PAOD) intended to be or treated by the VITUS peripheral drug-coated dilatation catheter when used according to the Instructions for Use and treating physician decision. Data will be collected in order to assess the long-term safety and performance of the VITUS peripheral drug-coated dilatation catheter in routine clinical practice.

DETAILED DESCRIPTION:
The multicenter, prospective registry population consists of consecutive patients with peripheral arterial occlusive disease (PAOD) who undergo percutaneous transluminal angioplasty (PTA) intervention and are intended to be or treated by the VITUS peripheral drug-coated dilatation catheter (according to the Instructions for Use) as part of routine clinical care. Approximately 284 patients from approximately 15 centers in Europe will be entered into the registry. Patients entered into the registry are followed for three years. The registry is considered finished when all patients have completed the 36-month follow-up.

A follow-up is scheduled at the following timepoints: immediately post-procedure, 30 days, 6 months, 12 months, 24 months, and 36 months. Follow-up is obtained by telephone contact with the patient or at a planned hospital visit.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients intended to be or treated by the VITUS peripheral drug-coated dilatation catheter as per physicians' decision and according to IFU in the setting of routine clinical care are entered into the registry
* The lesion to be treated should be shorter than the nominal length of balloon at a reference vessel diameter of 2.0 mm up to 7.0 mm.

  * If lesion is longer than the individual balloon, more than one DCB can be used for longer lesions with the mandatory overlapping balloons of 10mm to avoid any geographical miss.
* Rutherford clinical categories 2-5

Exclusion Criteria:

* The patients are excluded from registration if ANY of the following conditions apply:

  * High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
  * Currently participating in another investigational drug or device study in which a routine angiographic follow-up in peripheral arteries is planned
  * A life expectancy of <1year
  * Explicit refusal of participation in the registry
  * Residual stenosis >50% after vessel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic peripheral arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 284 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Adjudicated freedom from major adverse events (MAE) | 30 days post-procedure (primary safety endpoint at 30 days)
  Adjudicated freedom from major adverse events (MAE), where MAE is defined as a composite of device- and procedure-related mortality, freedom from major target limb amputation, and freedom from clinically driven target lesion revascularization (cd-TLR)
Proportion of participants with Adjudicated freedom from major adverse events (MAE) | 12 months post-procedure (primary safety and efficacy endpoint at 12 months)
  Adjudicated freedom from MAE, where MAE is defined as a composite of device- and procedure-related mortality through 30 days, freedom from major target limb amputation, and freedom from clinically driven target lesion revascularization (cd-TLR) within 12 months
Occurrence of Adjudicated freedom from cd-TLR | 12 months post-procedure (primary efficacy endpoint at 12 months)
  Adjudicated freedom from cd-TLR, where cd-TLR is defined as any reintervention performed for ≥50% diameter stenosis (visual estimate) at the target lesion after documentation of recurrent clinical symptoms

SECONDARY OUTCOMES:
Proportion of participants with Adjudicated freedom from MAE | 6 months
  Adjudicated freedom from MAE, where MAE is defined as a composite of device- and procedure-related mortality through 30 days, freedom from major target limb amputation, and freedom from clinically driven target lesion revascularization (cd-TLR) within 6 months
Occurrence of Adjudicated freedom from cd-TLR | through hospital discharge (expected to be within 24 hours), at 30 days, 6 months, 24 months and 36 months
  Adjudicated freedom from clinically driven target lesion revascularization (cd-TLR)
Occurrence of Adjudicated freedom from clinically driven target vessel revascularization (cd-TVR) | through hospital discharge (expected to be within 24 hours), at 30 days, 6 months, 12 months, 24 months and 36 months
  Adjudicated freedom from clinically driven target vessel revascularization (cd-TVR)
Proportion of participants with Major amputation-free survival | through hospital discharge (expected to be within 24 hours), at 30 days, 6 months, 12 months, 24 months and 36 months
  Major amputation-free survival, defined as absence of target limb major amputation (above the ankle)
Proportion of participants with Any amputation-free survival | through hospital discharge (expected to be within 24 hours), at 30 days, 6 months, 12 months, 24 months and 36 months
  Any amputation-free survival, defined as absence of any amputation in target limb
Proportion of participants with Adjudicated freedom from MAE | through hospital discharge (expected to be within 24 hours), 6 months, 12 months, 24 months and 36 months
  Adjudicated freedom from MAE
Change in Rutherford clinical category | 12 months
  Mean change in rate from baseline Rutherford clinical category (clinical assessment at hospital visit)
Change in Walking Impairment Questionnaire (WIQ) results | 12 months, 24 months, and 36 months
  Mean change in rate from baseline in Walking Impairment Questionnaire (WIQ) results (telephone interview questionnaire)
Proportion of participants with Primary patency | 12 months, 24 months, and 36 months
  Primary patency, defined as freedom from >50% restenosis in the target lesion as indicated by a peak systolic velocity ratio >2.4 on duplex ultrasound or by visual assessment of an angiogram (if patients visit hospital), or freedom from clinically-driven reintervention (if telephone contact)
Proportion of participants with Device Success | Peri-procedural
  Device Success: Successful reaching of the target lesion, inflation and deflation of the balloon catheter, and a final residual stenosis after DCB treatment of ≤30% by visual assessment
Proportion of participants with Procedure Success | Peri-procedural
  Procedure Success: Successful balloon delivery, deployment, and retrieval, with no peri-procedural death, or target vessel revascularization (TVR)
Quality of Life Assessment | 12 months
  Mean change from baseline in European Quality of Life-5 Dimensions (EQ-5D) questionnaire The descriptive system assesses the quality of life and has one question for each of the five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. These answers are combined and converted to an index with 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Principal Investigator — AZ St Blasius Dendermonde
Locations (12):
- Belgium (6):
  - AZORG, Aalst
  - AZ Sint-Blasius, Dendermonde
  - ZOL Genk, Genk
  - AZ Groennge, Kortrijk
  - RZ Heilig Hart Tienen, Tienen
  - AZ Jan Portaels, Vilvoorde
- Germany (2):
  - Klinikum Lippe Detmold, Detmold
  - SRH Klinikum Karlsbad-Langensteinbach GmbH, Karlsbad
- Spain (4):
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital General de Granollers, Granollers
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario de Toledo, Toledo

IPD SHARING:
Plan to Share IPD: No